CLINICAL TRIAL: NCT00983502
Title: Pilot Study of Alternative Treatments of Unexplained Chronic Fatigue
Status: Terminated | Type: Observational
Why Stopped: IRB ended and NIH study ended
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 25988; R21AT004537-02 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Idiopathic Chronic Fatigue; Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Idiopathic Chronic Fatigue; Chronic Fatigue Syndrome; Myalgic encephalomyelitis
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Integrative Medicine: Patients of MD practitioners trained in Complementary and Alternative Medicine
- Naturopath Doctors: Patients of practitioners who are not MD's and are trained in Naturopathic Medicine
- Chronic Fatigue Specialists: Patients of MD's who specialize in treating Chronic Fatigue and related conditions
- Control Group: Patients treated by primary care MDs in practice-based research networks

SUMMARY:
The investigators' long-term goal is to identify, and then provide general practitioners with evidence-based recommendations for therapeutic interventions for unexplained chronic fatigue (UCF). The investigators' central hypothesis guiding this application is that some complimentary and alternative medicine (CAM) practitioners have developed management approaches that are more helpful to patients with UCF than usual care.

DETAILED DESCRIPTION:
An objective is to identify certain types of clinicians (or individual physicians) who appear to have identified effective treatments for patients with UCF, or to find that clinicians who report themselves to be effective are not. Study subjects will be UCF patients new to the practice of one of four groups of participating clinicians: 1) a control group of MDs in practice-based research networks, 2) MDs trained in CAM, 3) naturopathic doctors (non MDs trained in special naturopathic schools), and 4) MDs who specialize in chronic fatigue. Our rationale for this comparison is that its successful completion will potentially guide future searches for effective medical strategies for the treatment of UCF that may have been developed outside the mainstream medical community. It may also provide necessary information for follow-up studies that will help to identify specific effective treatments. This information includes which clinicians provide the best treatments (as evidenced by having patients with the best results), what are the characteristics of patients who respond to a particular treatment, how the data collection procedures might need to be refined and what sample sizes are necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 through 65.
2. Has severe debilitating fatigue that substantially reduces the quality of life.
3. Does not have any organic, psychological, or lifestyle problems that are the primary disorder and are likely to be the cause of this fatigue (see exclusionary criteria)
4. The severe, unexplained fatigue has persisted for at least six months.
5. Has not been previously treated by current physician for chronic fatigue.
6. Can speak and read English.
7. Is not pregnant or planning to become pregnant within six months.
8. Has a telephone.

Exclusion Criteria:

No known history of:

1. Bipolar disorder
2. Psychosis
3. Major Depressive Disorder
4. Sleep disorder
5. Anemia
6. Thyroid disease
7. Rheumatoid Arthritis
8. Systemic Lupus
9. Cancer
10. Heart disease
11. Liver disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The primary analyses will compare outcomes for 240 patients in four main groups (60 in each group) defined by the background of the treating clinicians. Study subjects will be UCF patients new to the practice of one of four groups of participating clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Differences among four groups of clinicians with respect to patient treatment outcome | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Hartz, MD, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States